CLINICAL TRIAL: NCT07383428
Title: IGHID 12601 - Improving Neurodevelopment With an Intestinal Health and Caregivers' Intervention in the surOeste, Guatemala: The INICIO-Guatemala Study
Brief Title: The INICIO-Guatemala Study
Acronym: INICIO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 26-0089; R01HD116306 (NIH)
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Development, Child
Keywords: Nutritional intervention; Microbiome; Caregiving; Rice bran; Bean flour

STUDY DESIGN:
Intervention Model Description: 2x2
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nutritional Intervention (Experimental): Children in this arm will receive the Nutri-INICIO intervention between 6 and 24 months of age.
  Interventions: Dietary Supplement: Nutri-INICIO
- Caregiver Intervention (Experimental): Caregivers of child participants in this arm will be trained in the Mediational Intervention for Sensitizing Caregivers (MISC) between 12 and 24 months of child age.
  Interventions: Behavioral: Mediational Intervention for Sensitizing Caregivers (MISC
- Nutritional Intervention and Caregiver Intervention (Experimental): Children in this arm will receive the Nutri-INICIO intervention between 6 and 24 months of age and their caregivers will be trained in the MISC between 12 and 24 months of child age.
  Interventions: Dietary Supplement: Nutri-INICIO; Behavioral: Mediational Intervention for Sensitizing Caregivers (MISC
- Active Control (Active Comparator): Children in this arm will receive the same number of study visits as the experimental groups and will receive essential components of the Minister of Health's childcare package, including micronutrient supplementation.
  Interventions: Other: Active Control

INTERVENTIONS:
Dietary Supplement: Nutri-INICIO — Nutri-INICIO, is a fortified maize-bean-rice bran porridge intended to improve intestinal health and growth. Caregivers will be instructed on Nutri-INICIO preparation methods. Children 6-11 months old will receive a 20 gram daily serving, children 12-17 months old will receive a 30 gram daily serving, children 18-24 months old will receive a 40 gram daily serving. The investigators will ensure receipt of the essential components of the ministry of health childcare package including micronutrient supplementation and anti-parasite prophylaxis. Participants will also receive anemia screening and treatment as appropriate.
  Arms: Nutritional Intervention; Nutritional Intervention and Caregiver Intervention
Behavioral: Mediational Intervention for Sensitizing Caregivers (MISC — The Mediational Intervention for Sensitizing Caregivers (MISC) consists of twice-monthly, video-feedback-based training sessions from 12-24 months to enhance responsive caregiving. The investigators will ensure receipt of the essential components of the ministry of health childcare package including micronutrient supplementation and anti-parasite prophylaxis. Participants will also receive anemia screening and treatment as appropriate.
  Arms: Caregiver Intervention; Nutritional Intervention and Caregiver Intervention
Other: Active Control — The control group will receive the same number of visits as the experimental groups and the investigators will ensure receipt of the essential components of the ministry of health childcare package including micronutrient supplementation and anti-parasite prophylaxis. Participants will also receive anemia screening and treatment as appropriate.
  Arms: Active Control

SUMMARY:
The goal of this randomized controlled trial (RCT) is to evaluate an intestinal health-targeted nutritional intervention and a caregiver training program, individually and combined, on childhood neurodevelopment (ND) in rural southwest Guatemala.

The main questions it aims to answer are: what is the impact of an intestinal-targeted nutritional intervention on child ND and what is the added benefit of a caregiver intervention on child ND.

The primary endpoint is the Mullen Scales of Early Learning (MSEL) Early Learning Composite (ELC) Score at 24 months. Secondary endpoints include MSEL subdomain scores (gross motor, fine motor, expressive language, receptive language, visual reception).

Researchers will compare child ND between the four study arms using a factorial design: (1) intestinal health-targeted nutritional intervention, (2) caregiving training program, (3) combined intestinal health-targeted nutritional intervention and caregiving training program, and (4) active control.

Participants will be randomized as mother-child dyads at 6 months of age and followed until 24 months of age.

DETAILED DESCRIPTION:
The investigators plan to enroll 400 pregnant women during the second trimester of pregnancy; randomization of mother-child dyads into the four study groups will occur at 6 months of infant age; infants will be followed through 24 months of age. Randomization will occur using a 2×2 factorial design into the four groups. The nutritional intervention, Nutri-INICIO, is a fortified maize-bean-rice bran porridge intended to improve intestinal health and growth. The caregiver intervention, the Mediational Intervention for Sensitizing Caregivers (MISC), consists of twice-monthly, video-feedback-based training sessions from 12-24 months to enhance responsive caregiving.

ELIGIBILITY:
The investigators will offer enrollment to pregnant in the Trifinio region of southwest Guatemala and will enroll their newborns after birth.

Inclusion Criteria:

* Pregnant woman in the second trimester of pregnancy
* Pregnant woman =>15 years of age
* Plan to live in the study area during pregnancy and up to 24 months after giving birth
* Newborns born to enrolled women will join the study at birth

Exclusion Criteria:

* Pregnant woman less than 15 years of age
* Planning to move during the study
* Not willing or able to participate in the interventions, including following instructions for preparing the food, completing the adherence forms, participating in the caregiving sessions
* Women who do not sign the consent form for their or their child's participation
* Infants who require a hospital stay after birth of 21 days or longer

Ages: 0 Days to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-06-15 (Estimated); Primary Completion 2030-06-15 (Estimated); Study Completion 2030-06-15 (Estimated)

PRIMARY OUTCOMES:
Mullen Scales of Early Learning (MSEL) Early Learning Composite Score (ELC) | 24 months of age
  Comprehensive neurodevelopment score, combining scores from the four "cognitive" domains of fine motor, visual reception, receptive language, and expressive language. Z-scores for each of the 4 domains will be calculated by regressing raw score for age. The mean of those four Z-scores will make up the Early Learning Composite Z-score. The score will range from -3 to +3, with the higher score indicating more advanced neurodevelopment.

SECONDARY OUTCOMES:
Mullen Scales of Early Learning Gross Motor Domain | 24 months
  The MSEL gross motor domain measures the child's gross motor development. A Z-score will calculated by regressing raw score for age. The score will range from -3 to +3, with the higher score indicating more advanced gross motor development.
Mullen Scales of Early Learning Fine Motor Domain | 24 months
  The MSEL fine motor domain measures the child's find motor development. A Z-score will calculated by regressing raw score for age. The score will range from -3 to +3, with the higher score indicating more advanced fine motor development.
Mullen Scales of Early Learning Visual Reception Domain | 24 months
  The MSEL visual reception domain measures the child's find motor development. A Z-score will calculated by regressing raw score for age. The score will range from -3 to +3, with the higher score indicating more advanced fine motor development.
Mullen Scales of Early Learning Receptive Language Domain | 24 months
  The MSEL receptive language domain measures the child's find motor development. A Z-score will calculated by regressing raw score for age. The score will range from -3 to +3, with the higher score indicating more advanced receptive language development.
Mullen Scales of Early Learning Expressive Language Domain | 24 months
  The MSEL expressive language domain measures the child's find motor development. A Z-score will calculated by regressing raw score for age. The score will range from -3 to +3, with the higher score indicating more advanced expressive language development.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Becker-Dreps, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Amy K Connery, PsyD, Principal Investigator — University of Colorado School of Medicine; Diva Mirella Barrientos Giron, MD, Principal Investigator — Fundacion para la Salud Integral de los Guatemaltecos
Locations (1):
- Fundacion para la Salud Integral de los Guatemaltecos, Coatepeque, Departamento de Quetzaltenango, Guatemala

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared at the time of publication. The data from this study will be made publicly available on the NICHD Data and Specimen Hub (DASH) (https://dash.nichd.nih.gov/) .
Time Frame: At the time of publication and will continue to be available for a period of at least 7 years.
Access Criteria: The data from this study will be made publicly available on the NICHD Data and Specimen Hub (DASH) (https://dash.nichd.nih.gov/).